CLINICAL TRIAL: NCT04167878
Title: 3D Printed Biodegradable Cervical Interbody Fusion Cage in Anterior Cervical Discectomy and Fusion，a Small Sample and Exploratory Research
Brief Title: Exploratory Study of 3D Printed Biodegradable Cervical Interbody Fusion Cage
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20192002-F-2
Record Dates: First submitted 2019-11-08; First posted 2019-11-19 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-06

CONDITIONS: Symptomatic Cervical Disc Disease

STUDY DESIGN:
Intervention Model Description: A total of 5 couple， 10 patients will be assigned into investigational (n=5) and control groups (n=5).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACDF with 3D printed biodegradable cervical fusion cage (Experimental): A resorbable cervical interbody cage made of PCL-TCP.
  Interventions: Device: 3D printed biodegradable cervical fusion cage
- ACDF with PEEK cage (Active Comparator): A structural PEEK cage with autologous bone.
  Interventions: Device: PEEK cage

INTERVENTIONS:
Device: 3D printed biodegradable cervical fusion cage — ACDF with 3D printed biodegradable cervical interbody fusion cage for spinal fusion procedure at one level (C2 to T1) of the cervical spine.
  Other Names: 3D printed PCL-TCP cage
  Arms: ACDF with 3D printed biodegradable cervical fusion cage
Device: PEEK cage — ACDF with PEEK cage for spinal fusion procedure at one level (C2 to T1) of the cervical spine.
  Arms: ACDF with PEEK cage

SUMMARY:
A small sample, single center, non-randomized, noninferiority clinical trial to evaluate the safety and effectiveness of 3D printed biodegradable cervical interbody fusion cage in anterior cervical discectomy and fusion (ACDF) for treating patients with a symptomatic degenerative cervical disc disease at one level from C2/C4 to C7/T1.

DETAILED DESCRIPTION:
The study will evaluate if 3D printed biodegradable cervical interbody fusion cage is non-inferior to poly-ether-ether-ketone (PEEK) cage in single-level ACDF with the use of local autologous bone. 3D printed biodegradable cervical interbody fusion cage is a restorable cervical interbody cage for the treatment of fusion, following discectomy, of the cervical spine from C2/C4 disc space to the C7/T1 disc space. The material used to prepare the implant is a mixture of polycaprolactone (PCL) and tricalcium phosphate (TCP), which is called PCL-TCP. The implant has proper strength and connective porosity. The PCL-TCP cage is intended to be used with a supplemental fixation system.

ELIGIBILITY:
Inclusion Criteria:

1. Skeletally mature patients aged between 25 and 85 years (inclusive);
2. Symptomatic cervical disc disease (SCDD) in the vertebral level between C2/C3 to C7/T1, correlated with radiculopathy or myelopathy;
3. Radiographic confirmation (by CT, MRI, x-ray, etc.) of any of the following: herniated nucleus pulposus, spondylosis or loss of disc height;
4. Requires only one cervical vertebral level to be surgically treated;
5. Failed at least 12 weeks of conservative treatment;
6. Patient must understand and sign the Informed Consent document that has been approved by the Ethics committee;
7. No significant restrictions showed by the pre-surgical routine test and examination.

Exclusion Criteria:

1. Skeletally immature patients;
2. Prior radiation history at anterior cervical area;
3. Prior surgery at the level to be treated;
4. More than one vertebral level requiring treatment, confirmed radiologically by X-ray, CT, or MRI
5. Complication of ossification of the ligamentum flavum, and Ossification of the posterior longitudinal ligament;
6. Clinically compromised vertebral bodies at the affected level(s) due to trauma or tuberculosis
7. Severe osteoporosis;
8. Active systemic or local infection;
9. Participation in other investigational device or drug clinical trials within 3 months of surgery;
10. Other patients whom the investigator believe not appropriate.

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Radiologic evaluation | 12 months
  Radiologic fusion assessed by roentgenographic examination or CT scan

SECONDARY OUTCOMES:
Japanese Orthopaedic Association Scores (JOA scores) | 12 months
  The whole name is Japanese Orthopaedic Association Scores for Assessment of Cervical spondylosis, the range of JOA is 0-17 and the full score is 17 to represent a normal function.
Measurement of Pain: Visual Analog Scale (VAS) | 12 months
  The whole name is Visual Analog Scale which is ranged from 0-10, with 0 being the least and 10 being the worst pain experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Guo, doctor, Principal Investigator — Department of orthopedics， Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China